CLINICAL TRIAL: NCT06722196
Title: BiodEgradable Soaked Amiodarone paTch Use for the Prevention of Atrial Fibrillation After Cardiac Surgery
Acronym: BEAT-AF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jilin Heart Hospital (Other)
Collaborators: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Jilin Heart Hospital 2024
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): patients will receive 2 patches soaked in cordarone hydrochloride (150 mg/3 ml each)
- Sham (Sham Comparator): patients will receive 2 patches soaked in saline solution (3 ml each)

INTERVENTIONS:
Drug: topical amiodarone — amiodarone soaked patch placed on the left atrial roof at the end of surgery
Other: saline solution patch — saline solution soaked patch placed on left atrial roof at the end of surgery

SUMMARY:
The primary objective of the present prospective, randomized, double blind, controlled study is to assess whether the application of 2 oxidized regenerated cellulose (SurgicelTM FibrillarTM) patches soaked with amiodarone hydrochloride over the anterior wall of the left atrium and the lateral wall of the right atrium results in a reduction in the incidence of POAF

ELIGIBILITY:
Inclusion Criteria:

* All patients who are candidates for elective cardiac surgery trough complete sternotomy with indications of coronary artery disease (both off-pump and on-pump), aortic valve disease, mitral valve disease, tricuspid valve disease, and ascending aorta disease, whether as an isolated pathology or in combination

Exclusion Criteria:

* patients with a clinical history of atrial or ventricular arrhythmia of any nature and duration, patients undergoing reoperation, patients with emergency surgical indications due to acute myocardial infarction or cardiogenic shock, patients with thyroid disfunction, patients with HOCM and those with pacemakers or ICDs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
postoperative atrial fibrillation versus control | within 5 days after surgery
  incidence of in-hospital atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Massimo G Lemma, PhD, Principal Investigator — Jilin Heart Hospital
Locations (1):
- Jilin Heart Hospital, Changchun, Jinlin, China

IPD SHARING:
Plan to Share IPD: No